CLINICAL TRIAL: NCT02597075
Title: Physical Activity in Patients With Metastatic Colorectal Cancer Who Receive Palliative First-line Chemotherapy. A Multicenter Open Label Randomized Controlled Trial
Brief Title: Physical Activity in Patients With Metastatic Colorectal Cancer Who Receive Palliative First-line Chemotherapy
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Feasibility (low patient accrual and financial reasons)
Sponsor: Swiss Cancer Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SAKK 41/14 - ACTIVE-2; 2015-003733-10 (EudraCT Number); 2015-003733-10 (Other: SNCTP)
Record Dates: First submitted 2015-10-22; First posted 2015-11-04 (Estimated); Last update posted 2022-11-07 (Actual); Status verified 2022-11

CONDITIONS: Metastatic Colorectal Cancer
Keywords: Colorectal Cancer; Metastatic Colorectal Cancer; Physical Activity; Quality of life
MeSH Terms: conditions — Colorectal Neoplasms; Motor Activity | interventions — Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm A: with ST + PA (Active Comparator): Standard therapy + structured Physical activity and pedometer
  Interventions: Other: standard therapy + physical activity program
- Arm B: (Active Comparator): Standard therapy
  Interventions: Other: standard therapy

INTERVENTIONS:
Other: standard therapy + physical activity program
  Arms: Arm A: with ST + PA
Other: standard therapy
  Arms: Arm B:

SUMMARY:
The purpose of this study is to assess whether a structured physical activity program (PA) during palliative chemotherapy improves progression-free survival (PFS) and/or patient-reported outcomes (ESAS-r) in patients with metastatic colorectal cancer.

DETAILED DESCRIPTION:
While safety and feasibility as well as some improvements in fitness, fatigue and certain aspects of quality of life have been shown for physical activity in cancer patients during treatment, none of the pre-requisites above (i-iv) is fulfilled in the setting of patients with advanced colon cancer.

However, evidence, primarily from the adjuvant setting, that physical activity impacts on treatment tolerability and tumor progression is a strong enough rationale to now embark on this prospective trial. By assessing in a large randomized controlled trial whether a 12-week structured physical activity program during chemotherapy in patients with newly diagnosed colorectal cancer undergoing standard first-line chemotherapy improves progression-free survival as compared to standard first-line chemotherapy alone, all pre-requisites for a practice-changing intervention are met.

The physical exercise ACTIVE-program describes a 12-week exercise program consisting of a combination of a bi-weekly aerobic exercise (cycle ergometer) supervised by a physical therapist and a self-paced increase in physical activity during daily life using a pedometer with a daily step goal as a motivational tool.

In addition to the supervised exercise program twice a week, patients of the intervention group are recommended to be physically active at home.

All patients will undergo standard systemic therapy for metastatic colorectal cancer. Patients in the care-as-usual group are not actively encouraged to change their physical activity level e.g. to start a fitness program during chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent according to ICH/GCP regulations before randomization.
* Patient with histologically or cytologically confirmed colorectal carcinoma (CRC) who start palliative first-line systemic therapy for inoperable or metastatic disease.

Note: Patients can be included before the start or within the first three weeks of first-line systemic treatment.

* Patients with histologically or cytologically confirmed colorectal carcinoma (CRC), who start first-line "conversion"-therapy for borderline resectable metastatic disease and will be reassessed for metastasectomy after 3-4 months of systemic treatment.

Note: Patients can be included before the start or within the first three weeks of first-line systemic treatment.

Patients who are diagnosed with metastatic disease and were initially treated with surgery and/or radiochemotherapy to the primary tumor are eligible (except if all disease sites/metastases have been removed) Patients who have been curatively treated with histologically or cytologically confirmed nonmetastatic CRC previously and now relapse with metastatic disease are also eligible, irrespective of previous radiochemotherapy and/or adjuvant chemotherapy

* Patients must have measurable disease on CT scan or MRI to be performed within 6 weeks before randomization (measurability criteria according to RECIST 1.1, non-nodal lesions ≥10 mm, lymph nodes ≥15mm) OR evaluable disease i.e. patient with nonmeasurable metastases but elevated serum tumor-marker (CEA at least >2xULN).
* Command of written and spoken language allowing for informed consent and for filling in trial questionnaires.
* Baseline patient-reported outcomes (PROs) have been completed.
* WHO performance status 0-2.
* Age ≥18 years

Exclusion Criteria:

* Pre-existing severe medical conditions precluding participation in a physical activity program as determined by the local investigator. Such conditions include: chronic heart failure (greater than NYHA II), recent myocardial infarction (less than 3 months ago), unstable angina pectoris, clinically significant arrhythmias, uncontrolled hypertension with repeated systolic blood pressure above 160mmHg, and COPD (requiring oxygen supply or GOLD stadium greater than 2).
* Inability to ride a cycle ergometer e.g. for musculoskeletal reasons.
* Patients in whom all CRC metastases have been removed surgically. It is allowed to include patients for whom metastasectomy might be an option if chemotherapy induces a significant response.
* Any serious underlying medical condition (at the judgment of the investigator) which could impair the ability of the patient to participate in the trial (e.g. active autoimmune disease, uncontrolled diabetes).
* Concurrent treatment in a trial with experimental drugs or other anti-cancer therapy, which are hypothesized to alter tumor progression. Participation in an observational trial or a translational trial is allowed. Palliative radiotherapy is allowed.
* Psychiatric disorder precluding understanding of trial information, giving informed consent, filling out PRO forms, or interfering with compliance.
* Any psychological, familial, sociological or geographical condition potentially hampering proper compliance with the trial protocol.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2016-03-17 (Actual); Primary Completion 2021-09-21 (Actual); Study Completion 2021-11-30 (Actual)

PRIMARY OUTCOMES:
Progression-free survival (PFS) | every 8 or 9 weeks during one year
  Change between 2 tumor assessments
Change in Patient-reported symptoms as measured by ESAS-r | in at week 6, 12, 18, 24, 48
  The ESAS-r is a summary score ranging from 0 to 100 with lower scores representing better quality of life of the patients.

SECONDARY OUTCOMES:
Overall survival | after progression (expected 1 year) lifelong follow-up
  time from randomization to date of death. Patients without event at the time of analysis will be censored at the date they were last known to be alive.
Best Objective Response | at week 8 or 9 during one year
  best tumor response achieved during first-line systemic therapy according to RECIST criteria. Only remission status achieved during first-line therapy will be considered.
Selected adverse events | day 1 of each cycle (every 8 or 9 weeks)
  assessed according to NCI CTCAE v4.0.
Chemotherapy-completion-rate | week 6, 12, 18, and 24
  total dose in mg which was applied divided by the total dose in mg which was initially planned according to the planned chemotherapy scheme. Absolute doses of chemotherapy agents applied will be collected after each chemotherapy cycle. The total planned dose will be derived based on the planned chemotherapy scheme which is specified at baseline incorporating weight or body surface.
  The chemotherapy-completion-rate is defined as the number of dose modifications due to toxicity during the first 24 weeks after randomization per patient: after each 6 week-period (week 6, 12, 18, and 24) it is assessed whether there have been dose modifications (decrease/delay of systemic treatment i.e. chemo or biological) due to toxicity during the previous 6 weeks (y/n). The proportion of patients without any dose modification due to toxicity during the first 24 weeks will be calculated as well
Initiation or increase of anti-hypertensive drugs | day 1 of each cycle (every 8 or 9 weeks) for one year
  In the subgroup of patients who receive bevacizumab. The proportion of patients receiving new or increased doses of anti-hypertensive drugs will be calculated.

CONTACTS AND LOCATIONS:
Overall Officials: Viviane Hess, Prof Dr med, Study Chair — University Hospital, Basel, Switzerland
Locations (24):
- Austria (2):
  - Universitätsklinikum der PMU Salzburg, Salzburg
  - Klinikum Wels-Grieskirchen GmbH, Wels
- Switzerland (22):
  - Tumor Zentrum Aarau, Aarau
  - Kantonsspital Aarau, Aarau
  - Kantonsspital Baden, Baden
  - St. Claraspital, Basel
  - Clinical Cancer Research Center at University Hospital Basel, Basel
  - Istituto Oncologico della Svizzera Italiana IOSI, Bellinzona
  - Spitalzentrum Biel, Biel
  - Spitalzentrum Oberwallis, Brig
  - Kantonsspital Graubünden, Chur
  - Hôpital Fribourgeois HFR, Fribourg
  - Hôpitaux Universitaires de Genève, Geneva
  - Centre de Chimiothérapie Anti-Cancéreuse, Lausanne
  - Kantonsspital Baselland, Liestal
  - Kantonsspital Luzern, Lucerne
  - Spital Thurgau, Münsterlingen
  - Kantonsspital Olten, Olten
  - Kantonsspital - St. Gallen, Sankt Gallen
  - SpitalSTS AG Simmental-Thun-Saanenland, Thun
  - Onkozentrum - Klinik im Park, Zurich
  - Onkozentrum Hirslanden Zürich, Zurich
  - Stadtspital Triemli, Zurich
  - UniversitätsSpital Zurich, Zurich

IPD SHARING:
Plan to Share IPD: No